CLINICAL TRIAL: NCT06640881
Title: Preoperative Partial Breast Reirradiation and Repeat Breast-conserving Surgery in Patients With Recurrent Breast Cancer: the REPEAT Trial - a Study Protocol
Brief Title: Preoperative Partial Breast Reirradiation and Repeat Breast-conserving Surgery in Patients With Recurrent Breast Cancer: the REPEAT Trial
Acronym: REPEAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Desiree H.J.G.D. van den Bongard, MD Ph, Dr, Principal Investigator, Radiation Oncologist, VU University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL85983.018.24
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Breast Carcinoma; Ipsilateral Recurrence
Keywords: single-dose preoperative radiotherapy; pathologic response; radiologic response; cosmetic outcome; partial breast irradiation
MeSH Terms: conditions — Breast Neoplasms | interventions — BaseLine dental cement; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ablative single-dose PBI followed by BCS after three weeks (Experimental): Eligible patients with a low-risk ipsilateral recurrent breast cancer previously treated with breast-conserving surgery and postoperative radiotherapy, will be treated with re-irradiation (i.e. ablative single-dose PBI) followed by second BCS after three weeks.
  Interventions: Radiation: ablative single-dose PBI

INTERVENTIONS:
Radiation: ablative single-dose PBI — ablative single-dose PBI followed by BCS after three weeks At baseline (prior to RT) and prior to BCS, toxicity, PROMS and cosmetic outcome will be assessed. Additionally, a preoperative MRI will be performed three weeks following RT to evaluate the acute tumor response.
  Other Names: baseline (prior to RT) and prior to BCS, toxicity, PROMS and cosmetic outcome will be assessed.; a preoperative MRI will be performed three weeks following RT to evaluate the acute tumor response

SUMMARY:
Over the past decades, interest in second breast-conserving therapy (BCT) has increased due to, among others, advancements in radiotherapy techniques. Preoperative partial breast irradiation (PBI) is an experimental treatment for patients with low-risk primary breast cancer. This approach can downstage the tumor, and may possibly reduce toxicity and improve cosmetic outcomes compared to postoperative radiotherapy. This study aims to evaluate the feasibility of single-dose preoperative PBI and second breast-conserving surgery (BCS) for patients with an ipsilateral recurrent breast event (IRBE) after previous BCT.

The REPEAT trial is a multicenter, prospective, single-arm trial investigating ablative single-dose preoperative PBI in patients with an IRBE. Eligible patients are ≥ 50 years, have a unifocal non-lobular invasive breast cancer ≤ 2 cm, Bloom-Richardson grade 1 or 2, estrogen receptor-positive, HER2-negative and clinically negative axillary lymph nodes. The study plans to enroll 25 patients. Radiotherapy planning will involve the use of CT and MRI in the treatment position. Single-dose PBI of 20 Gy to the tumor and 15 Gy to the surrounding 2 cm of breast tissue will be delivered using a conventional or MR-guided linear accelerator. Tumor response will be monitored preoperatively using MRI and liquid biopsies to identify biomarkers for evaluating radiosensitivity. BCS will be performed 3 weeks post-PBI. The primary endpoint is the incidence of grade 2 or higher treatment-associated acute toxicity within 90 days. Secondary endpoints include the evaluation of acute (grade 1) and late toxicity, radiologic and pathologic response, mastectomy rate, patient-reported outcomes, cosmetic outcome, local, regional and distant recurrence rates, survival outcome, and biomarkers in liquid biopsies and tumor tissue. Patients will be followed up to 5 years after PBI.

This trial will evaluate the feasibility of single-dose preoperative PBI and BCS for patients with IRBE. This treatment approach is expected to minimize the irradiated volume, reduce toxicity, and improve cosmetic outcomes compared to postoperative PBI after second BCS. Identifying biomarkers for radiosensitivity will help in selection patients and tailoring treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 50 years with an ipsilateral invasive recurrent breast cancer event after previous breast-conserving surgery and postoperative whole breast irradiation
* World Health Organization performance status 0-2
* Tumor size ≤ 2 cm and unifocal on MRI
* Tumor histology as assessed on biopsy:

Bloom-Richardson grade 1 or 2 Non-lobular invasive histological type carcinoma Estrogen receptor positive HER2 receptor negative No lymphovascular invasion

* No extensive DCIS (outside tumor size of 2 cm) on mammography or tumor biopsy, including non-mass enhancement on MRI
* Clinical node negative on 18-F FDG PET-CT, ultrasound and MRI
* No distant metastasis
* No or mild late toxicity (no grade 2 or higher) from previous breast-conserving therapy
* Adequate understanding of the Dutch language

Exclusion Criteria:

* Ipsilateral invasive breast cancer event less than two years after first breast-conserving therapy for breast cancer
* Other malignancy within 5 years before ipsilateral breast recurrence diagnosis. For carcinoma in situ no specific time span to ipsilateral breast recurrence diagnosis is required for inclusion
* Known breast cancer mutation gene carrier
* Collagen synthesis disease (e.g. osteogenesis imperfect, Ehlers-Danlos syndrome, systemic sclerosis)
* Previous ipsilateral mastectomy
* Invasive lobular carcinoma, DCIS without invasive cancer
* MRI absolute contraindications
* Indication for treatment with neoadjuvant chemotherapy
* Legal incapacity

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 90 days
  The incidence of grade 2 or higher treatment-associated acute toxicity within 90 days

SECONDARY OUTCOMES:
Toxicity | 3,6,12 weeks and 1,2,3,4,5 years
  Assessment of treatment-induced toxicity
response | 3,6,12 weeks and 1,2,3,4,5 years
  Assessment of radiologic and pathologic response, mastectomy rate
PROMS | 3,6,12 weeks and 1,2,3,4,5 years
  Assessment of PROMs
cosmetic results | 3,6,12 weeks and 1,2,3,4,5 years
  Assessment of cosmetic results
oncological outcomes | 1,2,3,4,5 years
  Assessment of oncological outcomes
immune response | 3,6,12 weeks and 1,2,3,4,5 years
  Assessment of RT-associated immune response and biomarkers in blood and tumor tissue
patient comfort during RT treatment delivery | during RT treatment
  Assessment of patient comfort during RT treatment delivery

CONTACTS AND LOCATIONS:
Overall Officials: Desiree HJG van den Bongard, dr, Principal Investigator — AUMC
Locations (1):
- Amsterdam UMC / VU Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Civil Y, Wurfbain L, Jonker L, van der Sangen M, Oei A, Duvivier K, Bijker N, Meijnen P, van Kesteren Z, Palacios M, Barbe E, Menke-van der Houven van Oordt W, Diepenhorst G, Thijssen V, Slotman B, Verhoeff J, Schipper RJ, van den Bongard D. Preoperative partial breast reirradiation and repeat breast-conserving surgery in patients with recurrent breast cancer: the prospective single-arm REPEAT trial - a study protocol. BMJ Open. 2025 Jul 18;15(7):e096510. doi: 10.1136/bmjopen-2024-096510. PMID 40681188